CLINICAL TRIAL: NCT00654719
Title: The Influence of Enteral Nutrition on Functional Status and Inflammatory Activation in Patients With Congestive Heart Failure and Cardiac Cachexia.
Brief Title: Enteral Nutrition in Congestive Heart Failure and Cardiac Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart and Lung Institute (Other)
Collaborators: Nutricia Research Fundation (Other)
Responsible Party: Iwona Wójcicka-Bartłomiejczyk, director, Nutricia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 372/2000
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Heart Failure; Cardiac Cachexia
Keywords: Heart failure; cachexia
MeSH Terms: conditions — Heart Failure; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NutriDrink (Active Comparator): Nutritional supplementation that contains 600 kcal/day: protein content 20 g, carbohydrates 72 g, fat 26 g
  Interventions: Dietary Supplement: NutriDrink
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NutriDrink — Nutritional supplementation that contains 600 kcal/day: protein content 20 g, carbohydrates 72 g, fat 26 g
  Arms: NutriDrink
Dietary Supplement: Placebo — Nutritional supplementation containing only 12 kcal/day
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the effects of a high caloric drink on weight and several other clinical markers including quality of life in patients with unintentional weight loss (cachexia) due to chronic heart failure.

DETAILED DESCRIPTION:
Cardiac cachexia has been shown to be powerful independent predictor of mortality in patients with congestive heart failure (CHF). Unlike starvation, cachectic CHF patients present with a decrease of muscles and/or fat tissue. This probably depends, at least in part, on the level of inflammatory activation. Theoretically, it seems clear that nutritional status has to be improved in cardiac cachexia. It has been suggested that inflammatory activation in CHF may be due to endotoxin translocation through the edematous gut wall. Elevated endotoxin levels have been found in patients with acutely decompensated CHF, but these levels normalized with diuretic treatment. This finding may be of utmost importance. From one side it underscores the need for aggressive diuretic treatment to prevent translocation, from another side however, it suggests potential area for enteral treatment. Enteral route of nutrition may be highly beneficial by diminishing bacterial translocation from guts and/or endotoxin transfer, finally resulting in lower inflammatory activation Numerous experimental studies display that enteral feeding reduces bacterial translocation, endotoxin absorption and positively modulates function of local immune tissue.

A search of the literature shows that very little is known about the effectiveness of nutritional support on functional performance in cachectic CHF patients and actually no reports concern the influence of enteral feeding on immune activation of cachectic CHF patients. Recent information of some links existing between leptin, which is increased in CHF, and inflammatory activation in this syndrome speculate on a functional role of leptin in immune activation in CHF. As leptin is one of the most important hormones in the regulation of body energy metabolism, we think it is reasonable to look also into enteral feeding -induced changes of leptin and concomitant fluctuations of plasma cytokines.

During the last 12 months we have been using nutritional support in cachectic patients with CHF as an adjunct to standard therapy. We were surprised by a significant functional improvement that we observed in many instances. As most of these patients were subjected to aggressive multi-drug diuretic therapy as well, it was impossible to appreciate the role of enteral nutrition in this respect. We think, these observations are worth verification in more controlled prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Signing of informed consent,
* Patient with either gender with actual signs or symptoms of congestive heart failure of any origin with NYHA class no less then III,
* Presence of cardiac cachexia as defined above,
* Duration of symptoms of congestive heart failure of at least 6 months,
* Ejection fraction assessed by echocardiography ≤30%,
* Nutritional support will be offered solely to patients with their pharmacological treatment firmly established for at least 30 days.

Exclusion Criteria:

* Acute decompensation with clinically evident pulmonary or abdominal congestion,
* Any situation (apart from congestive heart failure) that may affect absorption of nutrients from the gut,
* Presence of active gastritis or ulcer,
* Presence of cancer,
* Presence of thyreotoxicosis,
* Type I diabetes mellitus,
* Pancreatic insufficiency,
* Treatment with β-blockers,
* Clinically relevant liver disease with significantly elevated enzymes (ALAT or AspAT or ALP 4 times above normal according to local norms),
* Body mass index > 25,
* unstable angina pectoris or other acute coronary syndromes within last three months,
* Participation in any other studies,
* Signs of uncooperative attitude,
* Known HIV virus infection,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2001-04; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | 18 weeks
Quality of Life | 18 weeks

SECONDARY OUTCOMES:
Lean tissue content, total plus arms and legs separately, as assessed by dual X-ray absorptiometry (DEXA) | 18 weeks
Fat tissue content, total plus arms and legs separately, as assessed by dual X-ray absorptiometry (DEXA) | 18 weeks
Serum levels of inflammatory markers including tumor necrosis factor, its soluble receptors 1 and 2, and interleukin-6 | 18 weeks
Biochemistry markers including cholesterol, low density lipoprotein, high density lipoprotein | 18 weeks
Left ventricular ejection fraction as assessed by echocardiography | 18 weeks
Exercise testing using spiroergometry | 18 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Applied Cachexia Research, Department of Cardiology, Charité Medical School, Campus Virchow-Klinikum, Berlin, Germany
- Silesian Center for Heart Diseases, Zabrze, Poland

REFERENCES:
- [Background] Anker SD, Ponikowski P, Varney S, Chua TP, Clark AL, Webb-Peploe KM, Harrington D, Kox WJ, Poole-Wilson PA, Coats AJ. Wasting as independent risk factor for mortality in chronic heart failure. Lancet. 1997 Apr 12;349(9058):1050-3. doi: 10.1016/S0140-6736(96)07015-8. PMID 9107242
- [Background] Anker SD, Ponikowski PP, Clark AL, Leyva F, Rauchhaus M, Kemp M, Teixeira MM, Hellewell PG, Hooper J, Poole-Wilson PA, Coats AJ. Cytokines and neurohormones relating to body composition alterations in the wasting syndrome of chronic heart failure. Eur Heart J. 1999 May;20(9):683-93. doi: 10.1053/euhj.1998.1446. PMID 10208789
- [Background] Niebauer J, Volk HD, Kemp M, Dominguez M, Schumann RR, Rauchhaus M, Poole-Wilson PA, Coats AJ, Anker SD. Endotoxin and immune activation in chronic heart failure: a prospective cohort study. Lancet. 1999 May 29;353(9167):1838-42. doi: 10.1016/S0140-6736(98)09286-1. PMID 10359409
- [Background] Sax HC, Illig KA, Ryan CK, Hardy DJ. Low-dose enteral feeding is beneficial during total parenteral nutrition. Am J Surg. 1996 Jun;171(6):587-90. doi: 10.1016/s0002-9610(96)00039-6. PMID 8678205
- [Background] Kotani J, Usami M, Nomura H, Iso A, Kasahara H, Kuroda Y, Oyanagi H, Saitoh Y. Enteral nutrition prevents bacterial translocation but does not improve survival during acute pancreatitis. Arch Surg. 1999 Mar;134(3):287-92. doi: 10.1001/archsurg.134.3.287. PMID 10088570
- [Background] Guihot G, Merle V, Leborgne M, Pivert G, Corriol O, Brousse N, Ricour C, Colomb V. Enteral nutrition modifies gut-associated lymphoid tissue in rat regardless of the molecular form of nitrogen supply. J Pediatr Gastroenterol Nutr. 1997 Feb;24(2):153-61. doi: 10.1097/00005176-199702000-00008. PMID 9106101
- [Background] Heymsfield SB, Casper K. Congestive heart failure: clinical management by use of continuous nasoenteric feeding. Am J Clin Nutr. 1989 Sep;50(3):539-44. doi: 10.1093/ajcn/50.3.539. PMID 2505606
- [Background] Abel RM, Fischer JE, Buckley MJ, Barnett GO, Austen WG. Malnutrition in cardiac surgical patients. Results of a prospective, randomized evaluation of early postoperative parenteral nutrition. Arch Surg. 1976 Jan;111(1):45-50. doi: 10.1001/archsurg.1976.01360190047008. PMID 812456
- [Background] Otaki M. Surgical treatment of patients with cardiac cachexia. An analysis of factors affecting operative mortality. Chest. 1994 May;105(5):1347-51. doi: 10.1378/chest.105.5.1347. PMID 8181317
- [Background] Anker SD, Rauchhaus M. Insights into the pathogenesis of chronic heart failure: immune activation and cachexia. Curr Opin Cardiol. 1999 May;14(3):211-6. doi: 10.1097/00001573-199905000-00004. PMID 10358792
- [Background] Zhao SP, Zeng LH. Elevated plasma levels of tumor necrosis factor in chronic heart failure with cachexia. Int J Cardiol. 1997 Feb;58(3):257-61. doi: 10.1016/s0167-5273(96)02873-2. PMID 9076551
- [Background] Steele IC, Nugent AM, Maguire S, Hoper M, Campbell G, Halliday MI, Nicholls DP. Cytokine profile in chronic cardiac failure. Eur J Clin Invest. 1996 Nov;26(11):1018-22. doi: 10.1046/j.1365-2362.1996.2560587.x. PMID 8957209
- [Background] Anker SD, Chua TP, Ponikowski P, Harrington D, Swan JW, Kox WJ, Poole-Wilson PA, Coats AJ. Hormonal changes and catabolic/anabolic imbalance in chronic heart failure and their importance for cardiac cachexia. Circulation. 1997 Jul 15;96(2):526-34. doi: 10.1161/01.cir.96.2.526. PMID 9244221
- [Background] Toth MJ, Gottlieb SS, Goran MI, Fisher ML, Poehlman ET. Daily energy expenditure in free-living heart failure patients. Am J Physiol. 1997 Mar;272(3 Pt 1):E469-75. doi: 10.1152/ajpendo.1997.272.3.E469. PMID 9124554
- [Background] Leyva F, Anker SD, Egerer K, Stevenson JC, Kox WJ, Coats AJ. Hyperleptinaemia in chronic heart failure. Relationships with insulin. Eur Heart J. 1998 Oct;19(10):1547-51. doi: 10.1053/euhj.1998.1045. PMID 9820994
- [Background] Cohn JN, Levine TB, Olivari MT, Garberg V, Lura D, Francis GS, Simon AB, Rector T. Plasma norepinephrine as a guide to prognosis in patients with chronic congestive heart failure. N Engl J Med. 1984 Sep 27;311(13):819-23. doi: 10.1056/NEJM198409273111303. PMID 6382011
- [Background] Joseph J, Gilbert EM. The sympathetic nervous system in chronic heart failure. Prog Cardiovasc Dis. 1998 Jul-Aug;41(1 Suppl 1):9-16. doi: 10.1016/s0033-0620(98)80026-1. PMID 9715818
- [Background] Snitker S, Pratley RE, Nicolson M, Tataranni PA, Ravussin E. Relationship between muscle sympathetic nerve activity and plasma leptin concentration. Obes Res. 1997 Jul;5(4):338-40. doi: 10.1002/j.1550-8528.1997.tb00561.x. PMID 9285841
- [Background] Haynes WG, Morgan DA, Walsh SA, Mark AL, Sivitz WI. Receptor-mediated regional sympathetic nerve activation by leptin. J Clin Invest. 1997 Jul 15;100(2):270-8. doi: 10.1172/JCI119532. PMID 9218503
- [Background] Haynes WG, Sivitz WI, Morgan DA, Walsh SA, Mark AL. Sympathetic and cardiorenal actions of leptin. Hypertension. 1997 Sep;30(3 Pt 2):619-23. doi: 10.1161/01.hyp.30.3.619. PMID 9322991
- [Background] Santos-Alvarez J, Goberna R, Sanchez-Margalet V. Human leptin stimulates proliferation and activation of human circulating monocytes. Cell Immunol. 1999 May 25;194(1):6-11. doi: 10.1006/cimm.1999.1490. PMID 10357875
- [Background] Loffreda S, Yang SQ, Lin HZ, Karp CL, Brengman ML, Wang DJ, Klein AS, Bulkley GB, Bao C, Noble PW, Lane MD, Diehl AM. Leptin regulates proinflammatory immune responses. FASEB J. 1998 Jan;12(1):57-65. PMID 9438411
- [Background] Levy JR, LeGall-Salmon E, Santos M, Pandak WM, Stevens W. Effect of enteral versus parenteral nutrition on leptin gene expression and release into the circulation. Biochem Biophys Res Commun. 1997 Aug 8;237(1):98-102. doi: 10.1006/bbrc.1997.7086. PMID 9266837
- [Background] Paccagnella A, Calo MA, Caenaro G, Salandin V, Jus P, Simini G, Heymsfield SB. Cardiac cachexia: preoperative and postoperative nutrition management. JPEN J Parenter Enteral Nutr. 1994 Sep-Oct;18(5):409-16. doi: 10.1177/0148607194018005409. PMID 7815671
- [Derived] Rozentryt P, von Haehling S, Lainscak M, Nowak JU, Kalantar-Zadeh K, Polonski L, Anker SD. The effects of a high-caloric protein-rich oral nutritional supplement in patients with chronic heart failure and cachexia on quality of life, body composition, and inflammation markers: a randomized, double-blind pilot study. J Cachexia Sarcopenia Muscle. 2010 Sep;1(1):35-42. doi: 10.1007/s13539-010-0008-0. Epub 2010 Oct 26. PMID 21475692